CLINICAL TRIAL: NCT00303953
Title: Phase II Study of PXD101 (NSC-726630) in Relapsed and Refractory Aggressive B-Cell Lymphomas
Brief Title: PXD101 in Treating Patients With Relapsed or Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01096; NCI-2009-01096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000462614; S0520 (Other: Southwest Oncology Group); S0520 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — belinostat

ARMS (1):
- Arm I (Experimental): Patients will receive an infusion of PXD101 once a day for 5 days. Treatment may repeat every 3 weeks for up to 2 years. Some patients will also undergo core biopsy and blood collection for laboratory studies before and after treatment.
  After finishing treatment, patients will be evaluated every 3-6 months for up to 3 years.
  Interventions: Drug: belinostat

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101

SUMMARY:
This phase II trial is studying how well PXD101 works in treating patients with relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma. PXD101 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate response rate in patients with relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma treated with PXD101.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. II. Estimate the 6-month progression-free survival rate in patients treated with this drug.

TERTIARY OBJECTIVES:

I. Determine the major histocompatability complex of class II proteins (HLA-DR, -DP, -DQ), TUNEL, and CD8 infiltration status, by immunochemistry on paired pre- and post-treatment tumor samples, in the first 20 patients enrolled.

II. Measure CIITA and HLA-DR mRNA expression using quantitative reverse transcriptase-polymerase chain reaction and determine, preliminarily, the associations of these markers with progression-free survival.

III. Evaluate paired pre- and post-treatment peripheral blood mononuclear cells from patients for histone acetylation status and determine correlation with findings from duplicate experiments on pre- and post-needle core biopsies.

OUTLINE: This is a multicenter study.

Patients receive PXD101 IV over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Needle core biopsies and peripheral blood mononuclear cells are obtained from the first 20 patients pre- and post-treatment for biomarker correlative studies.

After completion of study treatment, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven (no needle aspirations or cytologies) aggressive B-cell non-Hodgkin's lymphoma (NHL), including 1 of the following histology subtypes:

  * Diffuse large cell NHL
  * Burkitt's or Burkitt-like NHL
  * Primary mediastinal NHL
* Relapsed or refractory disease
* Bidimensionally measurable disease
* Transformed NHL allowed
* Not eligible for stem cell transplantation (for patients registered to study at first relapse)
* No active CNS involvement by lymphoma
* Zubrod performance status 0-2
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count>=100,000/mm^3
* WBC >= 3,000/mm^3
* Creatinine < 2 times upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min
* No significant EKG abnormalities
* Bilirubin normal
* SGOT/SGPT < 2.5 times ULN (=< 5 times ULN if liver involvement)
* No long QT syndrome or marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of QTc interval > 500 msec)
* No other significant cardiovascular disease, including any of the following:

  * Unstable angina pectoris
  * Uncontrolled hypertension
  * Congestive heart failure related to primary cardiac disease
  * Any condition requiring anti-arrhythmic therapy
  * Ischemic or severe valvular heart disease
  * Myocardial infarction within the past 6 months
* No major surgery within 28 days prior to study entry
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent medication that may cause Torsades de Pointes (i.e., prolongation of the QT interval > 500 msec)
* At least 14 days since prior radiotherapy
* At least 2 weeks since prior valproic acid or any other histone deacetylase inhibitor
* No clinical evidence of any of the following:

  * Severe peripheral vascular disease
  * Diabetic ulcers or venous stasis ulcers
  * History of deep venous or arterial thrombosis within the past 3 months
* Radioimmunotherapy is considered a chemotherapy regimen
* Single-agent rituximab is not considered a chemotherapy regimen
* Standard salvage chemotherapy followed by autologous stem cell transplantation is considered 1 regimen
* No known AIDS or HIV-associated complex
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix
* At least 2 weeks since prior therapy and recovered
* No more than 5 prior chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bernstein, Principal Investigator — SWOG Cancer Research Network
Locations (123):
- United States (123):
  - Providence Hospital, Mobile, Alabama
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Marin General Hospital, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Highland Hospital, Rochester, New York
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - McLeod Regional Medical Center, Florence, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Southwest Oncology Group, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- PXD101: Only eligible patients were included in the analyses. Patients receive 1000 mg/m^2 IV PXD101 on days 1-5 of each 21-day cycle until disease progression.
Period: Overall Study
Arm/Group | PXD101
Started | 22
Eligible | 21
Eligible and Treated | 20
Completed | 3
Not Completed | 19
Not completed — Ineligible | 1
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 12
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | PXD101
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 68.9 [51.6 to 82.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assess Number of Patients Who Achieve Confirmed and Unconfirmed Complete Response (CR) or Partial Response (PR)
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the SPD for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: assessed at week 8, and every 3 months for 3 years
Population: All eligible patients who started treatment were included in assessing response estimates.
Measure: Number; unit: participants
Groups:
- PXD101: Patients receive 1000 mg/m^2 IV PXD101 on days 1-5 of each 21-day cycle until disease progression.
Arm/Group | PXD101
Number analyzed (Participants) | 20
participants
  Complete Response (CR) | 0
  Complete Response Unconfirmed (CRU) | 0
  Partial Response (PR) | 0
  No response | 20

2. Secondary Outcome: Overall Survival
Description: Measured from time of registration to death, or last contact date
Time Frame: assessed every 3 months for 3 years
Population: Only eligible patients were included in the analyses.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | PXD101
Number analyzed (Participants) | 20
years | 0.9 [0.2 to 2.3]

3. Secondary Outcome: Progression-free Survival
Description: Measured from date of registration to time of first documentation of progression or death, or last contact date. Progression is defined as a 50% increase in sum of products of greatest diameters (SPD) of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline; appearance of a new lesion/site; unequivocal progression of non-measurable disease in the opinion of the treating physician; death due to disease without prior documentation of progression.
Time Frame: assessed at week 8, then every 3 months for 3 years
Population: Only eligible patients were included in the analyses.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | PXD101
Number analyzed (Participants) | 20
years | 0.2 [0.1 to 0.3]

ADVERSE EVENTS:
Time Frame: After every cycle while on protocol treatment, for a maximum of 2 years
Arm/Group | PXD101
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXD101 (N=20)
Hemoglobin (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Platelets (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PXD101 (N=20)
Hemoglobin (Blood and lymphatic system disorders) | 7
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Pain - Abdomen NOS (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Edema: limb (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 1
Injection site reaction/extravasation changes (General disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 6
Alkaline phosphatase (Investigations) | 4
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 1
Creatinine (Investigations) | 4
Leukocytes (total WBC) (Investigations) | 2
Lymphopenia (Investigations) | 2
Metabolic/Laboratory-Other (Specify) (Investigations) | 2
Platelets (Investigations) | 5
Prolonged QTc interval (Investigations) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Neurology-Other (Specify) (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes/flushes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Phlebitis (including superficial thrombosis) (Vascular disorders) | 2
Vascular-Other (Specify) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less